CLINICAL TRIAL: NCT04853199
Title: Effectiveness of Quercetin In The Treatment of SARS-COV 2
Brief Title: Quercetin In The Treatment Of SARS-COV 2
Acronym: QUERCOV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, Professor, Hôpital Universitaire Sahloul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QUERCOV
Record Dates: First submitted 2021-04-18; First posted 2021-04-21 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: SARS (Severe Acute Respiratory Syndrome)
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Quercetin

STUDY DESIGN:
Intervention Model Description: a randomized double-blind study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quercetin group (Experimental): Each patient included, after signing the consent, will have a treatment for ten days: one tablet twice a day 30 minutes before the meal
  Interventions: Drug: Quercetin
- Placebo Group (Placebo Comparator): Each patient included, after signing the consent, will have a treatment for ten days: one tablet twice a day 30 minutes before the meal
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quercetin — Each patient should receive one tablet twice a day 30 minutes before the meal
  Arms: Quercetin group
Drug: Placebo — Each placebo capsule contains 150 mg of microcrystalline cellulose and 1.5 mg of magnesium stearate.
  Arms: Placebo Group

SUMMARY:
In 1937, Albert Szent-Gyorgyi received a Nobel Prize for discovering vitamin C and flavonoids, as well as for exploring their biochemical properties. Originally, he gave the flavonoids the name "vitamin P" because of their effectiveness in reducing the permeability of blood vessels. This name was abandoned when it was realized that these substances were not really vitamins.

Quercetin is extracted from a variety of plant sources, including the onion peel and the seeds and pods of Dimorphandra mollis, a legume tree native to South America.

Although we are far from knowing everything about quercetin, its antioxidant, anti-inflammatory, and antihistamine (antiallergic) properties have been observed in numerous in vitro and animal studies.

DETAILED DESCRIPTION:
Properties

* Anti-oxidant, vascular protector
* Inhibition of platelet aggregation, vasorelaxant , arterial relaxant
* Anti-hypertensive , especially by certain derivatives (quercetin-3-glucuronic acid)
* Nephroprotective in rats, protects against the nephrotoxicity of gentamicin
* Anticancer , with immunostimulatory activity and inducer of apoptosis, with activity on the shock proteins HSP (heat shock proteins) hsp27 and hsp70
* Antitumor activity against prostate cancer and certain breast cancer cells
* Prevention of cardiac toxicity from doxorubicin, with resveratrol
* Protection against gastric inflammation associated with Helicobacter pylori infection by activity on MAPK, BCL-2, BAX.
* Increases the antitoxic activity of the liver
* Pancreatic lipase inhibitor, potential action in weight gain
* Anti-inflammatory
* Anti-allergic, inhibition of mast cell degranulation, with a preventive effect, reduction of inflammation linked to eosinophils (such as isoquercitrin regulates the Th1 / Th2 balance
* Antiviral (dose-dependent reduction of infectivity, decreases intracellular replication)
* Inhibition of rhinovirus replication
* Influenza prophylaxis by quercetin or its derivatives (quercetin-3-O-α-L-rhamnopyranoside), opposes the pro-oxidant effects induced by the influenza virus, antioxidant therapy could be used to prevent serious complications associated with influenza
* In vitro inhibition of the penetration of the Ebola virus by quercetin-3-O-glucoside
* Antiviral activity against Zika virus, hepatitis B virus, hepatitis C, Epstein-Barr virus EBV and antitumor against human gastric carcinoma

ELIGIBILITY:
Inclusion Criteria:

* • Clinical score greater than 6

  * Patients with clinical symptoms less than 5 days old.
  * Men and women at least 40 years old, able and willing to give informed consent;
  * Any patient over the age of 18 with a CT scan in favor of COVID-19;
  * Ambulatory or hospitalized environment;
  * Patient with dyspnea or with a positive gait test;
  * The patient must have at least one of the following high risk criteria: 70 years or older, obesity (BMI ≥ 30 kg / m2), diabetes mellitus, uncontrolled hypertension (systolic blood pressure ≥ 150 mm Hg), respiratory disease known (including asthma or chronic obstructive pulmonary disease), known heart failure, known coronary artery disease, fever ≥ 38.4 ° C within the last 48 hours, dyspnea at the time of presentation, bicytopenia, pancytopenia or a combination of a number high neutrophils and low lymphocytes count;
  * The patient is not of childbearing age, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing age and uses at least one method of contraception and preferably two complementary forms of contraception comprising a method of barrier throughout the study and for 30 days after the end of the study;
  * The patient must be able and willing to comply with the requirements of this study protocol.

Exclusion Criteria:

* • Patient currently in shock or exhibiting hemodynamic instability;

  * Patient with inflammatory bowel disease (Crohn's disease or ulcerative colitis), chronic diarrhea or malabsorption;
  * Pregnant or breastfeeding patient
  * Patient with a history of allergic reaction or significant sensitivity to Nigella;
  * The patient is considered by the investigator, for whatever reason, to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 30 days
  death rate
Need for ICU admission | 30 days
  Number of participants admitted to the Intensive care unit (ICU)
treatment safety | 30 days
  rate of adverse events

SECONDARY OUTCOMES:
Need for hospitalization for patients followed up at home | 30 days
  Need for hospitalization for patients followed up initially at home
lenghth of stay in Hospital | 30 days
  days spent at hospital for patients followed up initially at home
resolution of COVID-19 symptoms | 30 days
  Time to resolution of COVID-19 symptoms [ Evaluated at day 15 and day 30 precising the Time at which the patient is completely symptom free and severity of symptoms
need for oxygen therapy | 30 days
  Number of participants who needed oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukef, professor, Principal Investigator — CHU Sahloul, Sousse, Tunisia
Locations (2):
- Tunisia (2):
  - HU Sahloul, sousse, Tunisia, Sousse, Itinéraire Ceinture Cité Sahloul
  - Riadh Boukef, Sahloul, Sousse Governorate

IPD SHARING:
Plan to Share IPD: No
Two study groups will be included: 100 patients in the herbal medicine group and 100 patients in the Placebo group.
  For each patient included in the study, a PCR test for the detection of SARS-COV2 was performed with the prescription of a prescription containing: antibiotic therapy, paracetamol, cough syrup, mineral and vitamin supplements.
  A follow-up will be carried out for each patient included in the study every two days to note the clinical signs present and to verify compliance and adverse events for each.
  Data is entered on SPSS 21.0